CLINICAL TRIAL: NCT01532362
Title: Evaluation of Apricoxib (Selective Cyclooxygenase 2 Inhibition) in Modulating T Regulatory Cells of Patients With Early Stage Non-small Cell Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Drug sponsor stopped drug manufacture due to toxicity issues from other studies
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-002081
Record Dates: First submitted 2011-11-30; First posted 2012-02-14 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2013-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apricoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apricoxib (Experimental): As part of the trial, forty eligible subjects will be randomly assigned to receive Apricoxib 400 mg orally once daily or no drug intervention for a 7 day period (Days 0-6) prior to surgical resection of the lung tumor but between the two surgeries.
  Interventions: Drug: Apricoxib
- No drug intervention (Other)
  Interventions: Drug: Apricoxib

INTERVENTIONS:
Drug: Apricoxib — As part of the trial, forty eligible subjects will be randomly assigned to receive Apricoxib 400 mg orally once daily or no drug intervention for a 7 day period (Days 0-6) prior to surgical resection of the lung tumor but between the two surgeries.

SUMMARY:
The primary objective for this trial is to determine the biological ability of apricoxib to decrease T reg cells in the peripheral blood and tumor infiltrating lymphocytes in subjects compared to those who have not in subjects with early stage Non-small Cell Lung Cancer (NSCLC). The secondary objectives are to determine the efficacy of apricoxib to inhibit CD4+CD25+ T reg and FOXP3 function and exploration of COX-2 dependent biomarkers of apoptosis resistance, angiogenesis, invasion, and immunity.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 capable of giving informed consent. Radiographic findings suspicious for primary lung cancer or pathologically confirmed NSCLC which is surgically resectable and radiographically early stage (stage I and II).
* ECOG performance status of 0, 1, or 2 (see Appendix A).
* Ineligible for or refuse preoperative chemotherapy or chemoradiation therapy
* Normal renal function (defined as serum creatinine ≤ 2 mg/dl or creatinine clearance ≥ 60 ml/min/1.73m2).
* Normal liver function (defined as total bilirubin ≤ 1.5 x ULN, SGOT & SGPT ≤ 2.5 xULN).
* Negative pregnancy test prior to initiation of treatment and adequate contraception throughout treatment.
* Preoperative pulmonary function test (PFT) with FEV1 and D LCO ≥ 60% or predicted postoperative FEV1 and DLCO ≥ 40% based on quantitative lung perfusion scan
* Must be able to come off anticoagulants and have normal coagulation studies (PTT < 40 seconds and INR < 1.4) prior to planned surgery.
* For subjects on COX-2 inhibitors or other NSAIDS prior to study initiation, cessation of the drug for 1 week prior to Apricoxib administration is required for study enrollment.

Exclusion Criteria:

* Radiation therapy, chemotherapy, non-cytotoxic investigational agents, or corticosteroids within 4 weeks of initiating treatment.
* Comorbid disease or a medical condition that would impair the ability of the subject to receive or comply with the study protocol.
* Hypersensitivity to apricoxib, sulfonamides, aspirin, or other NSAIDS or to any reagents used in the study.
* Previous history of gastrointestinal ulceration, bleeding, or perforation.
* Required concurrent use of COX-2 inhibitors or other NSAIDS during Apricoxib administration.
* Chronic or concurrent use of steroids (topical steroids are acceptable if medically indicated).
* Pregnant or nursing women.
* Evidence of NYHA class III or greater cardiac disease.
* History of myocardial infarction, stroke, ventricular arrhythmia, or symptomatic conduction abnormality within 12 months of initiating treatment.
* History of heart surgery for coronary artery disease.
* Known HIV infection or AIDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay M Lee, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- No Drug Intervention: no drug intervention for a 7 day period (Days 0-6) prior to surgical resection of the lung tumor but between the two surgeries.
Period: Overall Study
Arm/Group | Apricoxib | No Drug Intervention
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: the truncated study had only one participant and that participant was on the Apricoxib arm of the study. Therefore the no drug intervention arm of the study had zero participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Apricoxib | No Drug Intervention | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Compare Level of CD4+CD25high T Lymphocyte Regulatory Cells in Peripheral Blood Lymphocytes and Tumor Infiltrating Lymphocytes From Surgical Resection Specimens of Subjects With Early Stage NSCLC Who Have Received Apricoxib to Those Who Have Not
Description: As part of the trial, forty eligible subjects will be randomly assigned to receive Apricoxib 400 mg orally once daily or no drug intervention for a 7 day period (Days 0-6) prior to surgical resection of the lung tumor but between the two surgeries. Peripheral blood and urine will be obtained on Days 0 and 7 from both groups (prior to surgical incision). Bronchoalveolar lavage (BAL) and lymph node tissue will be obtained on Days 0 and 7. TIL will be obtained from surgical resection specimens of the primary lung tumor only on Day 7
Time Frame: 7 days
Population: No analysis occurred
Arm/Group | Apricoxib | No Drug Intervention
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Effect of Apricoxib on Levels of CD4+CD25+ T Regulatory Cells in Peripheral Blood.Also,Biomarkers of Apoptosis Resistance,Angiogenesis,Invasion and Immunity Will be Tested in the Lab to Check How Effective Apricoxib is in Inhibiting These Proteins.
Description: Peripheral blood from patients with NSCLC has been reported to have an increase in the percentages of CD4+CD25+ T reg cells.In contrast <10% of the PBLs of normal donors have this phenotype. As such, CD4+CD25+ cells will be assessed in addition to FOXP3 levels in PBL. In addition, exploration of COX-2 dependent biomarkers of apoptosis resistance, angiogenesis, invasion, and immunity will be studied. COX-2, FOXP3, IL-10, IL-12, MDC, CXCR4 and survivin will be analyzed in plasma.
Time Frame: 7 days
Population: There was only one enrollee in this study. There was no analysis.
Arm/Group | Apricoxib | No Drug Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: from enrollment up to approximately 6 months
Description: There were no patients in the second arm of the study therefore the number of patients at risk of Adverse Events, Serious Adverse Events and All-Cause Mortality in that arm is zero.
Arm/Group | Apricoxib | No Drug Intervention
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Early termination of study when sponsor withdrew drug from market due to toxicities revealed from other studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No